CLINICAL TRIAL: NCT00067899
Title: Oxidative Stress and Vitamin E Requirements
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Maret Traber, Professor, National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: OSVER (completed)
Record Dates: First submitted 2003-08-29; First posted 2003-09-08 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Smoking
Keywords: cigarette smoking; tocopherol; bioavailability; metabolism; oxidative stress
MeSH Terms: conditions — Smoking; Cigarette Smoking | interventions — Vitamin E; Ascorbic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Vitamin E with and without Vitamin C

SUMMARY:
The purpose of this study is to determine if oxidative stress derived from cigarette smoking increases vitamin E requirements. The study will also assess the role of vitamin C in modulating vitamin E requirements. Vitamin E requirements will be assessed by measuring vitamin E in plasma as well as by measuring the excreted vitamin E metabolite in the urine.

DETAILED DESCRIPTION:
We will be investigating the fractional disappearance rate of tocopherols in cigarette smokers compared to nonsmokers. This will be accomplished by supplementing individuals with deuterium labeled alpha- and gamma-tocopherols. Quantification of plasma tocopherols as well as urinary metabolites, alpha- and gamma-carboxy ethyl hydroxychromanol, will be determined using liquid chromatography/mass spectrometry analysis. In addition, the role of vitamin C as it pertains to its influence on the fraction disappearance rate of vitamin E will also be evaluated.

ELIGIBILITY:
Inclusion criteria:

* non-smoking status or smokers (more than 1 pack per day)
* age: 18-35 y
* stable body weight, ranging between 80% and 130%,
* maintenance of normal exercise and activity patterns
* total cholesterol ≤ 7.758 mmol/L (300 mg/dl)
* triglyceride concentration ≤ 3.387 mmol/L (300 mg/dl)

Subjects will be excluded if they fulfill any one of the following:

* antioxidant supplement users
* resting blood pressure above 160/105 mm Hg
* engaged in aerobic activity more than five hours per week
* vegetarian or other restrictive dietary requirements
* fasting blood glucose concentration of ≥ 7.77 mmol/L (140 mg/dl)
* history of diabetes or uremia
* other known metabolic disease or medication use known to affect lipid metabolism

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 99
Dates: Start 2000-09; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Linus Pauling Institute - Oregon State University, Corvallis, Oregon, United States

REFERENCES:
- [Background] Traber MG, Winklhofer-Roob BM, Roob JM, Khoschsorur G, Aigner R, Cross C, Ramakrishnan R, Brigelius-Flohe R. Vitamin E kinetics in smokers and nonsmokers. Free Radic Biol Med. 2001 Dec 1;31(11):1368-74. doi: 10.1016/s0891-5849(01)00723-7. PMID 11728808
- [Background] Dietrich M, Block G, Norkus EP, Hudes M, Traber MG, Cross CE, Packer L. Smoking and exposure to environmental tobacco smoke decrease some plasma antioxidants and increase gamma-tocopherol in vivo after adjustment for dietary antioxidant intakes. Am J Clin Nutr. 2003 Jan;77(1):160-6. doi: 10.1093/ajcn/77.1.160. PMID 12499336
- [Background] Traber MG, van der Vliet A, Reznick AZ, Cross CE. Tobacco-related diseases. Is there a role for antioxidant micronutrient supplementation? Clin Chest Med. 2000 Mar;21(1):173-87, x. doi: 10.1016/s0272-5231(05)70016-2. PMID 10763098